CLINICAL TRIAL: NCT04114279
Title: Validation of a Totally Synthetic High Fidelity Laparoscopic Duodenal Atresia (DA) Surgical Simulator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jill Zalieckas, Associate in Surgery, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00032040
Record Dates: First submitted 2019-05-20; First posted 2019-10-03 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Duodenal Atresia
Keywords: surgical simulator
MeSH Terms: conditions — Familial duodenal atresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Duodenal Atresia Repair (Experimental): All participants will attempt a laparoscopic duodenal atresia repair on the synthetic high fidelity simulator.
  Interventions: Procedure: Performance of laparoscopic duodenal atresia repair

INTERVENTIONS:
Procedure: Performance of laparoscopic duodenal atresia repair — completion of laparoscopic duodenal atresia repair in a surgical simulator

SUMMARY:
Surgeons with variable levels of experience in pediatric minimally invasive surgery (MIS) will be recruited to test the laparoscopic DA simulator. Baseline characteristics regarding their experience level in pediatric surgery, open and laparoscopic DA repairs and MIS surgery will be obtained from all participants. Prior to testing the simulator, participants will be provided with a video and book chapter describing how to perform the procedures and will be given an opportunity to practice on the simulators. Participant performance during a DA repair will be video recorded. Their identity will be blinded. Time to completion will be recorded. Two expert assessors will score their performance using a checklist and global performance rating scale. The quality of the duodenal anastomosis will be scored. The performance of novice, intermediate and expert surgeons will be compared to determine if the DA simulator is able to distinguish between performance of surgeons at various levels of experience. In addition, post-procedure survey will be completed by participants to rate the simulators based on its realism, usability and usefulness. Recommendations for improvement to the simulator will be sought.

DETAILED DESCRIPTION:
All participants will be provided with chapters from a surgical atlas outlining the steps of a laparoscopic DA repair, as well as a video of a laparoscopic DA repair prior to testing the simulator. On the day of testing, they will also be given an opportunity to practice on the DA simulator. A pretesting survey will be completed to gather demographic information, surgical experience and self-reported comfort level at performing a laparoscopic DA repair. The survey responses will be used to stratify participants into experts (pediatric surgeons with ≥3 laparoscopic DA repairs and/or ≥5 advanced pediatric MIS procedures), intermediates (pediatric surgeons with <3 thoracoscopic TEF/EA repair or laparoscopic DA repairs and/or <5 advanced Pediatric MIS procedures) and novices (general surgeons or trainees without advanced Pediatric MIS experience) for analysis of results.

Participants will then be asked to perform a laparoscopic DA repair on the simulator. Their performance will be video recorded. Recordings include only the surgery being performed in the simulator, as a result there will be no identifying information in the recordings. Time to completion will be recorded. Two independent assessors will score the participants performance using the objective structured assessment tool (OSAT) global rating scale (GRS) and a task specific checklist. The repaired DA samples will be blinded and assessed for quality of anastomosis by scoring for completeness, patency, suture density, % of square knots, and leak pressures (see appendix 3).

Upon completion of the simulator testing a post-procedure survey will be completed by participants regarding their experience and to provide feedback on simulator.

ELIGIBILITY:
Inclusion Criteria:

* surgical resident with at least 3 years of training
* surgical critical care fellow
* pediatric surgery fellow
* pediatric surgery attending

Exclusion Criteria:

* surgery trainee with less than 3 years of training
* non-surgeon

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
1. Performance on the simulator as measured by a composite score of the OSAT (Objective Structured Assessment of Technical Skill) GRS (Global Rating Scale) and task specific checklist. | The OSAT and task specific checklists will be completed upon review of the videos by two blinded independent reviewers after all participants have completed simulator testing. It will be completed within one year of the study start date
  Participant operative performance based on OSAT GRS: There are 6 categories that are graded on scale of 1-5, where 5 is best performance. Categories include: respect for tissue, time&motion, instrument handling, flow of operation, knowledge of specific procedure, overall performance. A grade of 1-5 is given to each category.
  The task specific checklist ranks if the tasks involved in completion of procedure are 1. done correctly, 2. done incorrectly, 3. not done. There are 13 specific tasks for this procedure.
2. Realism of the DA simulator | The evaluation will be completed by participants immediately after performing the procedure.
  An evaluation of the trainer will be given to each participant upon completion of the procedure. The Evaluation includes a 5 point scale, where 5 is highly realistic, and 1 is unsure. The evaluation includes specific physical attributes of the trainer, realism of the materials, realism of the experience, ability to perform the specific tasks, and overall rating of the simulator. There is also a section for written comments
3. Utility of the simulator for teaching. | The evaluation will be completed by participants immediately after performing the procedure.
  The Evaluation form includes a section on the utility of the trainer as a training tool with a 5 point Likert scale - 5 being has great value and 1 being has no value
3. Utility of the simulator for assessment of skills. | The evaluation will be completed by participants immediately after performing the procedure.
  The Evaluation form includes a section on the utility of the trainer as a testing tool,with a 5 point Likert scale - 5 being has great value and 1 being has not value
3. Utility of the simulator for maintenance of skills | The evaluation will be completed by participants immediately after performing the procedure.
  The Evaluation form includes a section on the utility of the trainer as a tool for maintenance of skills,with a 5 point Likert scale - 5 being has great value and 1 being has no value

SECONDARY OUTCOMES:
1. Time to completion of the DA repair | On the day of simulator testing for each participant. We anticipate simulator testing to be completed within 6 months of the start date of the study.
  The time to completion of the DA repair will be recorded during simulator testing. It is defined by initial insertion of the instrument into the DA simulator to the time the participant cuts the final knot.
2. Anastomosis quality | Completed within 1 year of the start of the study
  Two blinded independent reviewers will review videos of procedures and the corresponding anastomosis specimen. They will rate the anastomosis quality based upon completeness (yes/no), patency (yes/no), suture density (length of incision and number of sutures - this is an evaluation of spacing of sutures. There is no optimal number, rather it is a balance of spacing appropriately to have enough sutures not to leak, but not too many, which will result in a prolonged procedure), % square knots (higher % is better), and leak pressures (high pressure is better).
3. Recommendations for improvement of the DA simulator | The evaluation will be completed by participants immediately after performing the procedure.
  Free text written feedback given by study participants on written section of evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Zalieckas, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No